CLINICAL TRIAL: NCT00024635
Title: The Evaluation of Patients With Mood and Anxiety Disorders and Healthy Volunteers
Brief Title: Evaluation of Patients With Mood and Anxiety Disorders and Healthy Volunteers
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: Suburban Hospital (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010254; 01-M-0254
Record Dates: First submitted 2001-09-23; First posted 2005-04-29 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-11-19

CONDITIONS: Mood Disorders; Anxiety Disorders; Healthy Volunteers; Bipolar Disorder; Depression
Keywords: Screening; Anxiety; Mood; Diagnostic Testing; Natural History
MeSH Terms: conditions — Mood Disorders; Anxiety Disorders; Bipolar Disorder; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Adult Healthy Volunteers: Adult Healthy Volunteers
- Adult Patients: Adult patients with mood and anxiety disorders
- Minor Healthy Volunteers: Minor Healthy Volunteers
- Minor Patients: Minor patients with mood and anxiety disorders
- Parents of Minor Healthy Volunteers: Parents and guardians of minor healthy volunteers
- Parents of Minor Patients: Parents and guardians of minor patients with mood and anxiety disorders

SUMMARY:
The purpose of this protocol is to allow for the careful screening of patients and healthy volunteers for participation in research protocols in the Experimental Therapeutics and Pathophysiology Lab (ETPB) at the National Institute of Mental Health (NIMH) and for the collection of natural history data. In addition the protocol will allow clinicians to gain more experience in the use of a variety of polysomnographic and high-density EEG recordings. Subjects in this protocol will undergo an evaluation which may include: a psychiatric interview; a diagnostic interview; rating scales; a medical history; a physical exam; brain magnetic resonance imaging (MRI); electroencephalography (EEG); electrocardiography (EKG), magnetoencephalography (MEG); blood, saliva and urine laboratory evaluation; and a request for medical records. Subjects may also be asked to complete questionnaires about attitudes towards research and motivation for research participation. The data collected may also be linked with data from other mood and anxiety disorder protocols (e.g., brain imaging, DNA, psychophysiology tests, treatment studies, etc) for the purposes of better understanding the diagnosis, pathophysiology, and treatment response of patients with mood disorders. Parents of minors will be interviewed. Upon conclusion of the screening process, subjects will either be offered participation in a research protocol and will sign the appropriate informed consent, or will be considered not appropriate for participation in research and will be referred back into the community. The current protocol thus serves as an entry point for individuals with mood or anxiety disorders or healthy volunteers to enter NIMH IRB approved ETPB protocols.

DETAILED DESCRIPTION:
The purpose of this protocol is to allow for the careful screening of patients and healthy volunteers for participation in research protocols on mood and anxiety disorders at the National Institute of Mental Health (NIMH) and for the collection of natural history data. Subjects in this protocol will undergo an evaluation which may include: a psychiatric interview; a diagnostic interview; rating scales; a medical history; a physical exam; brain magnetic resonance imaging (MRI); computed tomography (CT); electroencephalography (EEG); electrocardiography (EKG), magnetoencephalography (MEG); blood, saliva and urine laboratory evaluation; and a request for medical records. The data collected may also be linked with data from other mood and anxiety disorder protocols (e.g., brain imaging, DNA, psychophysiology tests, treatment studies, etc) for the purposes of better understanding the diagnosis, pathophysiology, and treatment response of patients with mood disorders. Parents of minors will be interviewed. Upon conclusion of the screening process, subjects will either be offered participation in a research protocol and will sign the appropriate informed consent, or will be considered not appropriate for participation in research and will be referred back into the community. The current protocol thus serves as an entry point for individuals with mood or anxiety disorders or healthy volunteers to enter NIMH IRB approved protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects ages 3 to 99 may enroll in the protocol.
* Subjects must be competent to comprehend the purpose of the screening process and to provide written informed consent and be willing to participate in NIMH IRB approved research protocols. Minors will be asked to assent and their parents will sign the consent form.
* Subjects will undergo an evaluation which may include a psychiatric interview, medical (including Tanner staging for minors), neurological, and laboratory examinations (as appropriate such as EKG, EEG, renal and liver function tests, serum electrolytes, urinalysis, HIV, hepatitis A, B, and C, lupus anticoagulant, anticardiolipin (aCL) antibodies, anti-b2glycoprotein-I antibodies, PT/PTT, blood levels of psychotropic drugs, pregnancy testing, and urine drug screen for the presence of psychoactive drugs and drugs of abuse).

EXCLUSION CRITERIA:

* Current alcohol or substance use or dependence (excluding nicotine) within the past 3 months of sufficient magnitude to require independent, concurrent treatment intervention (e.g. antabuse or opiate treatment, but not including self-help groups).
* Whether the minor lives with both parents or one parent, the parent(s) he/she lives with must have legal custody. If a parent has shared custody, both parents must consent to participate in this protocol.

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals being evaluated for mood and anxiety disorders and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2001-02-02 (Actual)

PRIMARY OUTCOMES:
Eligibility for research | Current and historical
  Evaluations of psychiatric and other medical conditions and histories to determine if the subjects are appropriate for participation in NIMH IRB approved protocols and for the collection of natural history data.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
During the screening process, if a clinical issue arises that warrants further evaluation and/or possible treatment, the subject will be informed and advised to seek medical care in the appropriate setting outside of NIH.

REFERENCES:
- [Derived] Ballard ED, Snider SL, Nugent AC, Luckenbaugh DA, Park L, Zarate CA Jr. Active suicidal ideation during clinical antidepressant trials. Psychiatry Res. 2017 Nov;257:303-308. doi: 10.1016/j.psychres.2017.07.065. Epub 2017 Jul 31. PMID 28787656
- [Derived] Nugent AC, Robinson SE, Coppola R, Zarate CA Jr. Preliminary differences in resting state MEG functional connectivity pre- and post-ketamine in major depressive disorder. Psychiatry Res Neuroimaging. 2016 Aug 30;254:56-66. doi: 10.1016/j.pscychresns.2016.06.006. Epub 2016 Jun 23. PMID 27362845
- [Derived] Ballard ED, Vande Voort JL, Bernert RA, Luckenbaugh DA, Richards EM, Niciu MJ, Furey ML, Duncan WC Jr, Zarate CA Jr. Nocturnal Wakefulness Is Associated With Next-Day Suicidal Ideation in Major Depressive Disorder and Bipolar Disorder. J Clin Psychiatry. 2016 Jun;77(6):825-31. doi: 10.4088/JCP.15m09943. PMID 27337418
- [Derived] Nugent AC, Iadarola ND, Miller FG, Luckenbaugh DA, Zarate CA Jr. Safety of research into severe and treatment-resistant mood disorders: analysis of outcome data from 12 years of clinical trials at the US National Institute of Mental Health. Lancet Psychiatry. 2016 May;3(5):436-42. doi: 10.1016/S2215-0366(16)00006-7. Epub 2016 Mar 10. PMID 26971192
- [Derived] Nugent AC, Robinson SE, Coppola R, Furey ML, Zarate CA Jr. Group differences in MEG-ICA derived resting state networks: Application to major depressive disorder. Neuroimage. 2015 Sep;118:1-12. doi: 10.1016/j.neuroimage.2015.05.051. Epub 2015 May 30. PMID 26032890
- [Derived] Machado-Vieira R, Yuan P, Brutsche N, DiazGranados N, Luckenbaugh D, Manji HK, Zarate CA Jr. Brain-derived neurotrophic factor and initial antidepressant response to an N-methyl-D-aspartate antagonist. J Clin Psychiatry. 2009 Dec;70(12):1662-6. doi: 10.4088/JCP.08m04659. Epub 2009 Sep 8. PMID 19744406
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2001-M-0254.html